CLINICAL TRIAL: NCT05701176
Title: A Clinical Imaging Study of the Changes in [18F]F-AraG Uptake Following Anti-PD-1 Therapy in Non-small Cell Lung Cancer
Acronym: SHARP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Idris Bahce, Idris Bahce, MD, PhD, Principal Investigator, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL78588.029.21
Record Dates: First submitted 2022-12-21; First posted 2023-01-27 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Advanced Stage Non-small Cell Lung Cancer
Keywords: Positron Emission Tomography; [18F]F-AraG; T-Lymphocytes; Longitudinal Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- [18F]F-AraG PET procedures (Experimental): All patients will undergo a total of 3 [18F]F-AraG PET scanning procedures at T=0, T=2 weeks and T=6 weeks.
  Interventions: Diagnostic Test: [18F]F-AraG PET scan

INTERVENTIONS:
Diagnostic Test: [18F]F-AraG PET scan — [18F]F-AraG PET scans are performed to assess the accumulation of activated T-cells in the tumour and healthy tissue.

SUMMARY:
[18F]F-AraG is a promising tracer to image activated T-cells with positron emission tomography (PET). The aim of the SHARP trial is to investigate changes in [18F]F-AraG uptake following Anti-PD-1 therapy in patients with non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
The efficacy of immunotherapy and patient selection for combinatorial immunotherapy strategies would greatly improve if the tumor microenvironment (TME) could be characterized more accurately. Positron emission tomography (PET) using tracers that target immune cell subsets may provide a non-invasive means to immune profile the TME. Imaging T-cells can help in identifying 'hot' tumors, or parts of the tumor mass that have high concentrations of tumor infiltrating T-cells and also provide information on its activation.

A promising tracer to image activated T-cells is [18F]F-AraG. Based on the hypothesis that [18F]F-AraG will accumulate in activated T-cells, it is expected that [18F]F-AraG and PET will enable to identify tumors and tumor areas with high concentrations of tumor infiltrating activated T-cells on pathological assessment.

In the SHARP trial, participants receive 3 longitudinal [18F]F-AraG PET scans during anti-PD-1 immunotherapy to explore the changes in uptake of [18F]F-AraG during the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed NSCLC, a histological biopsy is mandatory, negative for epidermal growth factor receptor (EGFR) and anaplastic lymphoma kinase (ALK) mutations
* Be willing to provide either archival biopsy or fresh biopsy at screening.
* Stage IIIB-IV patients that are planned to be treated with anti-PD-1 monotherapy
* High PD-L-1 expression (≥50% TPS)
* No prior systemic therapy for the treatment of cancer
* Be willing and able to provide written informed consent for the trial.
* Have a performance status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
* Be above 18 years of age on day of signing informed consent.

Exclusion Criteria:

* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of day 0. Inhaled or topical steroids, and adrenal replacement steroid >10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
* Untreated or symptomatic brain metastases
* Additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Active infection requiring systemic therapy.
* A history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Active Hepatitis B or C.
* Psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Patient is pregnant or breastfeeding or expecting to conceive within the projected duration of the trial, starting with the screening visit through 12 weeks after the last administration of [18F]F-AraG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
To assess the relative change in uptake of [18F]F-AraG in tumor lesions and lymphoid organs on anti-PD-1 treatment | six weeks
  To assess the changes in tracer uptake in all tumor lesions and lymphoid organs (lymph nodes, spleen) between baseline and after 2 and 6 weeks on-treatment per [18F]F-AraG PET scan.
To correlate baseline [18F]F-AraG uptake and tumor response to anti-PD-1 therapy | twelve weeks
  To correlate baseline tumor [18F]F-AraG uptake and objective response rate (ORR, defined as complete response (CR) and partial response (PR)) at 6 and 12 weeks.
To correlate the change in [18F]F-AraG uptake between baseline and on-treatment and tumor response to anti-PD-1 therapy | twelve weeks
  To correlate change in tumor [18F]F-AraG uptake as measured between baseline and 2 weeks and 6 weeks on-treatment, respectively, and objective response rate (ORR, defined as complete response (CR) and partial response (PR)) at 6 and 12 weeks.

SECONDARY OUTCOMES:
To assess the relationship between baseline tumor uptake of [18F]F-AraG, T cell infiltration and activation state at baseline | twelve weeks
  To correlate tumor [18F]F-AraG uptake at baseline with viable tumor cells and T-cell infiltration in tumor and stroma using multiplex IHC (VECTRA) analysis panels for T-cell subsets, for monocytes and metabolic milieu, and panels directed at resistance as well as RNA sequencing to assess tumor microenvironment.

OTHER OUTCOMES:
To assess the relationship between change of tumor uptake of [18F]F-AraG and changes in PBMC subsets | six weeks
  To correlate changes in tumor [18F]F-AraG uptake as measured between baseline and 2 weeks and 6 weeks on-treatment, with changes in the immune profile of peripheral blood mononuclear cells (PBMC) as measured between baseline and 2 weeks and 6 weeks on-treatment.
To visually correlate the [18F]F-AraG autoradiogram with immuno-histochemistry (IHC) read outs for tumor cells and T-cells | twelve weeks

CONTACTS AND LOCATIONS:
Overall Officials: Idris Bahce, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- Amsterdam UMC, location VU University Medical Center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No